CLINICAL TRIAL: NCT02456233
Title: Randomized Evaluation of Conventional Ablation With or Without Focal Impulse and Rotor Modulation to Eliminate Human Atrial Fibrillation (RECONFIRM): A Randomized Clinical Trial
Brief Title: Evaluation of Conventional Ablation With or Without Focal Impulse and Rotor Modulation to Eliminate Human AF
Acronym: RECONFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Director of AF Program and EP Research, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECONFIRM2015; K24HL103800 (NIH)
Record Dates: First submitted 2015-05-24; First posted 2015-05-28 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: rotor; FIRM; paroxysmal atrial fibrillation; persistent atrial fibrillation; atrial tachyarrhythmia; ablation; contact mapping; clinical trial; signal processing
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional AF Ablation with PVI (Active Comparator): These patients will be treated by conventional AF ablation by pulmonary vein isolation (PVI) alone.
  Interventions: Procedure: Conventional AF Ablation with PVI
- FIRM-guided ablation plus PVI (Experimental): These patients will be treated by ablation of patient-specific rotors and focal sources (FIRM). Conventional ablation (PVI) will then be performed as part of the standard of care procedure.
  Interventions: Procedure: FIRM-guided ablation plus PVI

INTERVENTIONS:
Procedure: Conventional AF Ablation with PVI — Trigger Based Ablation for AF, using Pulmonary Vein Isolation (PVI) alone
  Arms: Conventional AF Ablation with PVI
Procedure: FIRM-guided ablation plus PVI — Substrate ablation for AF, via ablation of rotors and focal sources. Conventional (PVI) ablation will also be performed.
  Arms: FIRM-guided ablation plus PVI

SUMMARY:
This prospective randomized study will assess the safety and efficacy of FIRM-guided ablation (FIRM+PVI) compared to pulmonary vein isolation (PVI) without FIRM, for the treatment of symptomatic atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) affects over 2 millions Americans. AF may reduce cardiac performance and may result in thrombus formation in the left atrium and thromboembolic events, such as stroke. Ablation to eliminate the causes of this arrhythmia is increasingly performed since pharmacological therapy is suboptimal. Ablation currently targets triggers, by ablating left atrial areas outside the pulmonary veins (pulmonary vein isolation, PVI) in subjects with symptomatic AF who have failed drugs. Unfortunately, this has mixed success with the best outcomes being 50-70% freedom from AF at 1 year post ablation.

A major issue with AF therapy is the lack of knowledge about critical regions of the heart that cause and sustain AF. A recent trial (STAR-AF2) showed that ablating regions empirically - i.e. without defining their role in AF(lines or fractionated electrograms) - did not improve patient outcomes compared to PVI alone (Verma et al, NEJM 2015). However, this leaves us with PVI that had a 50% success rate in that trial and in several other trials even for paroxysmal AF.

We hypothesize that guiding ablation to critical arrhythmia-targeting zones will improve success over PVI alone. Specifically, we hypothesize that computational mapping of AF will find small regions called rotors and focal sources and ablate them, called Focal Impulse and Rotor Modulation (FIRM) ablation, shows promise at eliminating AF substrates. In many single center trials, FIRM improves results from PVI alone. This will be among the first randomized comparisons of FIRM ablation compared to PVI alone, and addresses an important question in the field.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 years
2. Reported incidence of at least two documented episodes of symptomatic paroxysmal or persistent atrial fibrillation (AF) during the 3 months preceding trial entry (at least one episode documented by 12-lead ECG or ECG rhythm strip). Ideally, patients will have implanted continuous ECG recorders in place for >30 days prior to the procedure to document AF episodes and percentage of time in AF ("burden") prior to ablation
3. Male -or- Women without childbearing potential (surgically sterile or have been without a period for 12 months), -or- Women of childbearing potential who are not pregnant per a serum HCG lab test
4. Refractory to at least one Class I or III anti-arrhythmic medications. Drug doses must be therapeutic and stable
5. Willingness, ability and commitment to participate in baseline and follow-up evaluations without participation in another clinical trial (unless documented approval received from both sponsors)
6. Oral anticoagulation required for those subjects who have a score of two or more based on the following criteria (CHA2DS2VASc)

   * congestive heart failure (1 point)
   * hypertension (1 point)
   * age 75 years or older (2 points)
   * diabetes (1 point)
   * prior stroke or transient ischemic attack (2 points)
   * vascular disease (including coronary artery disease, CAD) (1 point)
   * age 65 years or older (1 point)
   * gender category: female (1 point) Pre-procedural anticoagulation will ideally have been continuous for 3 or more weeks prior to the procedure, as clinically indicated, with INR > 2 in patients taking warfarin.
7. Patient is willing and able to remain on anti-coagulation therapy for a minimum of 3 months post procedure for all subjects, and potentially indefinitely post procedure if the patient has CHA2DS2VASc score >or= 2
8. Signed, informed consent after a full discussion of the risks and benefits of both therapy arms, and the concept of randomization
9. NYHA Class 0, I or II and stable on medical therapy for > 3 months
10. Left atrial diameter <or= 5.5cm (CT or MRI preprocedure, or intracardiac echocardiography, with documented image of largest dimension)
11. LVEF >or= 40%
12. Sustained AF during procedure: If the patient does not experience spontaneous sustained AF (>10 min) during the procedure, typically in paroxysmal AF patients, sustained AF will be induced in routine fashion by burst pacing initially from the coronary sinus, then from other sites, then with isoproterenol infusion. Using intensive AF induction methods (Narayan, J Cardiovasc EP; 2012; 23(5): 447-454) sustained AF is induced in > 90% of paroxysmal AF patients presenting in sinus rhythm. If AF cannot be sustained, the patient does not meet the inclusion criteria for the protocol and the patient will undergo AF ablation per physician direction.

Exclusion Criteria:

1. Reversible Cause of Atrial Fibrillation: Atrial fibrillation from a reversible cause (e.g., surgery, hyperthyroidism, pericarditis); Cardiac or thoracic surgery (e.g., valve repair or coronary artery bypass grafting, CABG) within the last 180 days; AF secondary to electrolyte imbalance, thyroid disease
2. Anti-Coagulation Contraindicated: Contraindication to Heparin; Contraindication to Warfarin or other novel oral anticoagulants (e.g., dabigatran, rivaroxabanm apixaban); History of significant bleeding abnormalities
3. Clotting Diathesis: History of significant blood clotting abnormalities, systemic thrombi or systemic embolization
4. Cardiac Prosthesis: ASD closure device, LAA closure device, prosthetic mitral or tricuspid valve
5. Thrombus or Mass: Atrial clot/thrombus on imaging such as on a trans-esophageal echocardiogram (TEE) within 72 hours of the procedure; Intramural thrombus or other cardiac mass that may adversely affect catheter introduction or manipulation; Significant pulmonary embolus within 6 months of enrollment
6. Acute illness or active systemic infection or sepsis that may ordinarily warrant postponement of the procedure
7. History of recent cerebrovascular disease (stroke or TIA) or systemic thromboembolism within < 6 months
8. Severe Heart Failure: NYHA classes III, IV; Heart failure that is not stable on medical therapy; Pulmonary edema that may make planned anesthesia or sedation difficult
9. Non-Stable Coronary Disease: Stable/unstable angina or ongoing myocardial ischemia; Myocardial infarction (MI) within the past 3 months
10. Structural heart disease of clinical significance including:

    * Congenital heart disease where the abnormality or its correction prohibit or increase the risk of ablation
    * Acquired heart disease that may increase the risk of ablation, such as significant ventricular septal defect post myocardial infarction
    * Rheumatic valve disease, since this produces a unique AF phenotype
    * Extreme left atrial enlargement, defined as LA volume index > 60 ml/m2, in whom PVI has low success and 55 mm baskets are too small for the atria
11. Planned Cardiac Surgery: If cardiac transplantation or other cardiac surgery are planned within the 12 months follow period of the trial
12. Life expectancy less than 12 months (the followup period of the trial)
13. Significant pulmonary disease (e.g., COPD) or any other disease that significantly increase risk to the patient from sedation or anesthesia
14. Untreatable allergy to contrast media
15. Electrolyte imbalance: At the time of the ablation procedure, clinically significant abnormalities in serum potassium, sodium, magnesium or other electrolytes that affect the suitability of the patient for ablation at that time

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2025-02 (Actual); Study Completion 2025-02 (Actual)

PRIMARY OUTCOMES:
Long term success | 12 months
  Freedom from atrial fibrillation (AF) recurrence during the 12 months after the initial AF ablation procedure, after an initial 3 month blanking (healing and stabilization) period.

SECONDARY OUTCOMES:
Long-term freedom from AF/AT | 12 months
  Freedom from AF and atrial tachycardia (AT) during the 12 months after the initial AF ablation procedure, after an initial 3 month blanking (healing and stabilization) period. Atrial tachycardias (AT) include those arising from atrial regions where ablation was performed (such as left atrial tachycardia) as well as from regions where ablation was not performed (such as typical cavotricuspid isthmus dependent atrial flutter).
Total ablation time | 1 day
  Total ablation time will be recorded in all patients, measured as the cumulative application of energy from the first ablation lesion to the last lesion. These values will be compared between the FIRM-guided and conventional ablation groups. If ablation for AT/atrial flutter is pursued, this ablation time will be documented separately.
Quality of Life (comparing post-ablation to pre-ablation) | 12 months
  Quantitative EuroQol EQ5D scores post-ablation will be compared to those pre-ablation at all time points separately and together (ANOVA)
Adverse Events | 12 months
  Adverse events will be adjudicated by an independent Data and Safety Monitoring Committee, who will determine whether they are or are not related to the procedure. The number and type of adverse events will be compared between FIRM-guided and conventional ablation groups.
Healthcare Utilization | 12 months
  Hospitalization, other procedures and healthcare utilization, adjudicated by an independent Data and Safety Monitoring Committee, will be compared between limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Narayan, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center, San Diego, California
  - Stanford University, Stanford, California

REFERENCES:
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] Narayan SM, Baykaner T, Clopton P, Schricker A, Lalani GG, Krummen DE, Shivkumar K, Miller JM. Ablation of rotor and focal sources reduces late recurrence of atrial fibrillation compared with trigger ablation alone: extended follow-up of the CONFIRM trial (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation). J Am Coll Cardiol. 2014 May 6;63(17):1761-8. doi: 10.1016/j.jacc.2014.02.543. Epub 2014 Mar 13. PMID 24632280
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT02456233/ICF_000.pdf